CLINICAL TRIAL: NCT06203847
Title: A Randomized Clinical Trial of Patient Outcomes Following Out-of-Hospital Cardiac Arrest Receiving Epinephrine Versus In-together Vasopressin, Epinephrine, and Steroid. (OHCA REVIVES Trial)
Brief Title: The Effect of Prehospital Combination of Epinephrine, Vasopressin, and Steroid in OHCA
Acronym: REVIVES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 202204115MINA
Record Dates: First submitted 2023-12-18; First posted 2024-01-12 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Arrest; Out-Of-Hospital Cardiac Arrest; Emergency Medical Services
Keywords: Out-Of-Hospital Cardiac Arrest; Emergency Medical Services; Corticosteroid; Epinephrine; Vasopressin
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest; Diabetes Insipidus

STUDY DESIGN:
Intervention Model Description: a pragmatic randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant: adult patients with OHCA Outcomes Assessor: in-hospital care providers (physicians, nurses...etc)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Combined drug treatment: includes epinephrine (Adrenaline® 1mg/vial) every 3-5 minutes, vasopressin (Pitressin® 20Unints/vial) every 3-5 minutes up to 4 vials (a total of 80Units), methylprednisolone (Solu-Medrol® 40mg/vial).
  The method of administration is as follows: after the first administration of epinephrine (Adrenaline® 1mg/vial) to patients with cardiac arrest before hospital arrival, vasopressin (Pitressin® 20Unints/vial) and methylprednisolone (Solu-Medrol® 40mg/vial) are given simultaneously; thereafter, every 3-5 minutes, 1 mg (1 dose) of (Adrenaline® 1mg/vial) is given, along with 20 Units (1 dose) of vasopressin (Pitressin® 20Unints/vial) up to a maximum of 4 doses (a total of 80 Units) of vasopressin can be given before hospital arrival.
  Interventions: Drug: Combination group
- Control group (Active Comparator): Standard drug treatment: epinephrine (Adrenaline® 1mg/vial). According to international resuscitation guidelines ( Advanced Cardiac Life Support, ACLS), patients with cardiac arrest before hospital arrival are given 1 mg (1 dose) of epinephrine (Adrenaline® 1mg/vial) every 3-5 minutes.
  Interventions: Drug: Standard group

INTERVENTIONS:
Drug: Combination group — Combination of epinephrine (Adrenaline® 1mg/vial) every 3-5 minutes, vasopressin (Pitressin® 20Unints/vial) every 3-5 minutes up to 4 vials (a total of 80Units), methylprednisolone (Solu-Medrol® 40mg/vial)
  Arms: Intervention group
Drug: Standard group — standard doses of epinephrine (Adrenaline® 1mg/vial) every 3-5 minutes
  Arms: Control group

SUMMARY:
This project is a randomized controlled clinical research design, The hypothesis P-I-C-O of the study is: For adult patients in the Taipei City and New Taipei City communities who have suffered sudden non-traumatic death and have been resuscitated by advanced paramedics, the intervention group that receives combined drug treatment (epinephrine, vasopressin, methylprednisolone) has a better rate of sustained recovery of spontaneous circulation (ROSC) (primary outcome) and long-term survival status (secondary outcomes) compared to the control group that receives single drug treatment (epinephrine).

DETAILED DESCRIPTION:
The global and Taiwanese survival rates for patients following an out-of-hospital cardiac arrest (OHCA) are less than 10%. The emergency medical system (EMS) plays a crucial role in patient outcomes after OHCA, providing prehospital cardiopulmonary resuscitation, defibrillation, and medication. Among these medications, the combination of epinephrine, vasopressin, and methylprednisolone holds the most potential to improve patient survival rates following OHCA.

This study aims to compare the effect of standard epinephrine therapy with a combination of epinephrine, vasopressin, and methylprednisolone administered to OHCA patients. This comparison will be made through a randomized clinical trial (RCT) within the EMS of Taipei City and New Taipei City.

Throughout the research plan, we will conduct a prehospital RCT to answer the following question (in P-I-C-O format): Will adult non-traumatic OHCA patients resuscitated by paramedics in a prehospital setting have a better chance of sustained recovery of spontaneous circulation (primary outcome), and improved survival status (secondary outcomes), if they receive combination therapy (i.e., standard doses of epinephrine, 20U of vasopressin after each dose of epinephrine up to a maximum of 80U, and one dose of 40mg methylprednisolone after the first dose of epinephrine) compared to those who receive standard doses of epinephrine? We estimate a sample size of 1,344 OHCA patients to detect a difference in the primary outcome. Based on the background data from the EMS regions under study, we expect the enrollment to take approximately 30 months to complete.

This study is referred to as the "OHCA-REVIVES" trial, which stands for A randomized clinical trial of patient outcomes following Out-of-Hospital Cardiac Arrest Receiving Epinephrine Versus In-together Vasopressin, Epinephrine, and Steroid. The anticipated results from the "OHCA-REVIVES trial" will help determine the optimal strategy for prehospital medication, and will undoubtedly have a significant impact on resuscitation science. Through these efforts, we aim to improve the outcomes of OHCA patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged >= 18 )
* Out-of-hospital cardiac arrest in the studied regions
* Treated by paramedics authorized and capable of giving prehospital medication

Exclusion Criteria:

* OHCA with traumatic etiology
* Obvious signs of death like decapitation, rigor mortis, livor mortis, decomposition, etc.
* DNR (Do Not Resuscitation) or termination of resuscitation requested by the family
* Patients with known or suspected pregnancy
* No vascular access was established before hospital arrival
* ROSC before the administrated medication
* No patient contact (cancelled ambulance call or the patient was transported to the hospital before the arrival of trial-trained paramedics)
* Received epinephrine prior to the arrival of trial-trained paramedics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1344 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of sustained return of spontaneous circulation (ROSC) | estimated 2 hours
  Return of spontaneous circulation (ROSC) is the restart of a sustained heart rhythm measured by pulsation and vital signs that permeate the body after a cardiac arrest.
  Sustained ROSC ≥ 2 hours has been used as an surrogate to survival to hospital admission in many overcrowded emergency departments (ED).

SECONDARY OUTCOMES:
Rate of prehospital return of spontaneous circulation (ROSC) | estimated 1 hour
  presence of ROSC prior to arrival at emergency department (ED)
Rate of survival to hospital discharge | estimated 30 days
  survival to hospital admission, and without in-hospital death
Rate of survival with favorable neurologic status | estimated 30 days
  Good neurologic status (defined as Cerebral-Performance Category (CPC) score 1 and 2) at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: WEN CHU CHIANG, Phd, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study, the sharing of Individual Participant Data (IPD) will be made available in accordance with local privacy protection laws.
Supporting Information: Study Protocol
Time Frame: Upon completion of the study, estimated at the end of 2026, the sharing of Individual Participant Data (IPD) will be made available following local privacy protection laws.
Access Criteria: reasonable request to the corresponding authors.

REFERENCES:
- [Derived] Ko YC, Lin YY, Yang WS, Tseng YT, Huang TJ, Lai CT, Huang SY, Hsieh CM, Wang PL, Chen HH, Chen KY, Sun JT, Chang CH, Lu TP, Ma MH, Chiang WC. Vasopressin, steroids, and epinephrine in out-of-hospital cardiac arrest - a protocol for a randomized controlled trial (OHCA REVIVES trial). Resusc Plus. 2025 Nov 18;27:101163. doi: 10.1016/j.resplu.2025.101163. eCollection 2026 Jan. PMID 41399685